CLINICAL TRIAL: NCT03775278
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PHP-303 in Otherwise Healthy Overweight or Obese Subjects
Brief Title: A Study of Safety, Tolerability, and Pharmacokinetics of Multiple-Ascending Doses of PHP-303 in Otherwise Healthy Overweight or Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pH Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PHP-303-N102
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Otherwise Healthy Overweight or Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): PHP-303, multiple oral dose, up to 5 ascending dose cohorts
  Interventions: Drug: PHP-303
- Placebo (Placebo Comparator): Placebo, multiple oral dose, up to 5 ascending dose cohorts
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PHP-303 — Investigational drug
  Arms: Experimental
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled multiple-ascending dose (MAD) study designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of PHP-303 in otherwise healthy overweight or obese volunteer subjects. Within each ascending dose cohort, subjects will be randomized in a 4:1 ratio to receive PHP-303 or placebo. The primary objective is to establish the safety and tolerability and maximum tolerated dose (MTD) of orally-administered PHP-303.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ≥ 18 to ≤ 60 years of age.
* In good general health having no clinically significant diseases in medical history or evidence of clinically significant findings on physical examination, vital signs, laboratory results, and/or ECG at Screening, in the opinion of an Investigator.
* Willing to forego other forms of experimental treatment during the study.

Exclusion Criteria:

* Any clinically significant condition that, in the opinion of an Investigator, could preclude the safe participation of the subject in the study or would prevent the subject from meeting the study requirements.
* Major surgery in the 6 months preceding Screening.
* Clinically-significant abnormal laboratory parameters.
* Positive urine drug test for alcohol, cotinine, and/or drugs of abuse (cocaine, tetrahydrocannabinol, amphetamines, methamphetamines, or benzodiazepines) at Screening or on admission to the study site.
* Electrocardiographic Fridericia's corrected QT interval (QTcF) interval > 450 msec for males and > 470 msec for females, or any other clinically significant electrocardiographic abnormality.
* Blood pressure results > 150 mmHg systolic or > 95 mmHg diastolic
* Female subject who is pregnant (positive pregnancy test at the Screening Visit or on admission to the study site), lactating, or planning to become pregnant during the study period or within 3 months after the final dose of study medication.
* History of drug or alcohol abuse or dependence within 1 year prior to Screening.
* History of cigarette smoking within 3 months of Screening.
* Known intolerance to lactose.
* Regular use of prescription drugs within 14 days of the first administration of study drug or non-prescription (over-the-counter) drugs within 7 days of the first administration of study drug or unwilling to abstain from prohibited medications through the end of study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple oral doses of PHP-303 - Incidence of Adverse Events | Up to 12 weeks
  Assess the number of patients with adverse events
Safety and tolerability of multiple oral doses of PHP-303 - number of patients with abnormal ECG | Up to 12 weeks
  Number of patients with clinically significant change from baseline in standard 12 lead ECG parameters
Safety and tolerability of multiple oral doses of PHP-303 - blood pressure | Up to 12 weeks
  Number of patients with clinically significant change from baseline in systolic and diastolic blood pressure
Safety and tolerability of multiple oral doses of PHP-303 - heart rate | Up to 12 weeks
  Measured as number of heart beats per minute
Safety and tolerability of multiple oral doses of PHP-303 - body temperature | Up to 12 weeks
  Measurement of oral body temperature
Safety and tolerability of multiple oral doses of PHP-303 - respiratory rate | Up to 12 weeks
  Measured by number of breaths per minute
Plasma concentration of multiple oral doses of PHP-303 - AUC | Plasma Up to 12 weeks
  Area under the curve
Plasma concentration of multiple oral doses of PHP-303 - Cmax | Up to 12 weeks
  Maximum observed concentration
Plasma concentration of multiple oral doses of PHP-303 - Tmax | Up to 12 weeks
  Time to reach maximum measured plasma concentration
Plasma concentration of multiple oral doses of PHP-303 - t1/2 | Up to 12 weeks
  Determination of half-life

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Nicholls, MD, PhD, Study Chair — pH Pharma Inc
Locations (1):
- Vince & Associates Clinical Research, Inc., Overland Park, Kansas, United States